CLINICAL TRIAL: NCT04416906
Title: A Test and Treat Strategy in Barcelona: A Prospective Study in New HIV Diagnosis.
Brief Title: A Test and Treat Strategy in New HIV Diagnosis.
Acronym: Test&Treat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Judit Pich Martínez (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biktarvy Test&Treat; 2019-004837-17 (EudraCT Number)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm, single-centre prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biktarvy (Experimental): This is a fixed dose combination regimen containing 50 mg of Bictegravir + 200 mg of Emtricitabine + 25 mg of Tenofovir alafenamide.
  Interventions: Drug: Biktarvy

INTERVENTIONS:
Drug: Biktarvy — Once daily fixed dose combination regimen of Biktarvy will be evaluated as a rapid treatment strategy in newly HIV diagnosed patients HIV diagnosed patients that come for the first time to the Hospital Clínic HIV Unit

SUMMARY:
This is an open-label, single arm, single-centre prospective study to evaluate the feasibility, efficacy and safety of a once daily fixed dose combination regimen, Biktarvy, as a rapid treatment strategy in newly HIV diagnosed patients that come for the first time to the Hospital Clínic HIV Unit Patients with confirmed HIV-1 diagnosis who wish to start ARV treatment immediately will receive bictegravir 50 mg + emtricitabine 200 mg + tenofovir alafenamide 25 mg within the first week since the HIV-1 confirmation during 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Having confirmed HIV-1 positive test.
3. Patients not previously treated with antiretroviral treatment (post-exposure prophylaxis will be allowed if not done in the previous 6 months).
4. Clinically stable patients, in the opinion of the investigator, at the time of inclusion.
5. Women of child-bearing potential* must have a negative pregnancy test in urine before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: hormonal contraceptive methods intrauterine device, bilateral tubal occlusion, vasectomized partner or sexual abstinence.
6. Written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women at the time of the study inclusion or anticipating pregnancy during the follow-up period.
2. Suspicion of an active opportunistic infection that defers initiating antiretroviral treatment > 7 days since HIV confirmation.
3. Known hypersensitivity or intolerance of any of the components of Biktarvy®.
4. Patients on treatment with any prohibited medication (see section 5.2: Concomitant, nonpermitted and permitted medication).
5. Any condition which, in the opinion of the principal investigator, may interfere with adequate understanding, cooperation or compliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients non-eligible to receive any of the antiretroviral regimens within the first week since the HIV confirmation) at week 4 | week 4
  Patients will be considered non-eligible if they meet one or more of the following creiteria at week 4:
  * Presence of HLA-B* 5701 or lack of HLA test
  * Presence of HIV genotypic resistance mutations to at least one class of ARV drug that decrease efficacy of antiretroviral treatment
  * CD4 count < 200 cells/mm3
  * Viral load > 100.000 copies/mL
  * Comorbidities such as: Osteopenia measured by DXA (T score less than 1), medical history of cardiovascular risk measured by Framingham risk score > 10% at 10 years, Kidney function (eGFR <50mL/min),
  * Concomitant medication that can cause potential interactions with ARV (evaluating the risk of drug-drug interactions for drugs no totally safe (green colour) using the Liverpool website for DDI)
  * Hepatitis B (HBV) coinfection or lack of serology

SECONDARY OUTCOMES:
Proportion of patients who start Biktarvy within the first week since HIV confirmation at the first visit at the HIV unit. | week 4
Days since first HIV test was performed until Biktarvy is initiated. | week 4
Days since HIV confirmation (first visit at the HIV unit) until Biktarvy is initiated. | week 4
Proportion of patients with plasma viral load (VIH-1 RNA) < 50 copies/mL at 4, 12, 24 and 48 weeks. | week 4, week 12, week 24 and week 48
Changes from week 0 in CD4 and CD8 count and CD4/CD8 ratio at 24 and 48 weeks. | week 24 and week 48
Changes from baseline in systemic inflammatory and coagulation response evaluated by measurement of soluble markers including, but not limited to IL-6, ultrasensitive PCR, Dimer-D at 48 weeks. | week 48
Changes from baseline in senescence response evaluated by measurement of soluble markers of senescence including, but not limited to, bcl-2 apoptosis marker at 24 and 48 weeks. | week 24 and week 48
Proportion of patients who attend all the study visits (including blood collection) at 24 and 48 weeks. | week 24 and week 48
Changes from week 0 in subclinical obesity using dual x-ray absorptiometry at 48 weeks. | week 48
Proportion of patients with treatment-related adverse events during the study period. | week 48
Proportion of patients who discontinue study treatment due to adverse events at 48 weeks. | week 48
Changes in treatment adherence using the Simplified Medication Adherence Questionnaire at each visit during all the study period. | week 48
Patient perception of rapid start of Biktarvy therapy using a specific questionnaire (CESTA) at 48 weeks. | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Torres Berta, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
A plan description will be provided once it is decided

REFERENCES:
- [Derived] Ugarte A, De La Mora L, De Lazzari E, Chivite I, Fernandez E, Inciarte A, Laguno M, Ambrosioni J, Solbes E, Berrocal L, Gonzalez-Cordon A, Martinez-Rebollar M, Foncillas A, Calvo J, Blanco JL, Martinez E, Mallolas J, Torres B. Rapid initiation of bictegravir/emtricitabine/tenofovir alafenamide as first-line therapy in HIV infection. A prospective study. J Antimicrob Chemother. 2024 Sep 3;79(9):2343-2353. doi: 10.1093/jac/dkae235. PMID 39045754